CLINICAL TRIAL: NCT04274595
Title: Role of Reverse Transcriptase Inhibitors in the Treatment of Psoriasis: A Proof of Biological Concept Test
Brief Title: Role of Reverse Transcriptase Inhibitors in the Treatment of Psoriasis
Acronym: PSORTI-BIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOIGCSMerri/2018/PS-01; 2019-002236-91 (EudraCT Number)
Record Dates: First submitted 2020-01-16; First posted 2020-02-18 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psoriasis patients (Experimental)
  Interventions: Drug: Generic antiretroviral

INTERVENTIONS:
Drug: Generic antiretroviral — 200mg emtricitabine plus 245mg tenofovir diisopropyl fumarate for 7 days

SUMMARY:
The investigators hypothesize that the inhibition of endogenous reverse transcriptase would: (1) reduce excess cytosolic DNA, stress initiating the inflammatory loop at the origin of psoriatic lesions, and (2) interrupt the loop and lighten lesions

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from plaque psoriasis for more than a year with at least one active skin lesion> 4 cm2 in the photo-protected area.
* Patient using effective contraception (IUD, adapted pill, condom, etc.)
* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* Patient with another form or stage of psoriasis
* Patient on anti-cytokine treatment during the 6 months (180 days) before inclusion
* Patient under systemic treatment based on (1) corticosteroids, (2) antibiotics, (3) methotrexate, ciclosporin, soriatane, hydroxyurea, apremilast or (4) PUVA, (5) UVB, (6) vitamin D3 during the 4 weeks (28 days) before inclusion
* Patient on topical corticosteroid or retinoid treatment during the 2 weeks (15 days) before inclusion
* Patient with renal insufficiency; taking nephrotoxic agents (aminoglycosides, multiple or high doses of NSAIDs, etc.); creatinine clearance less than 50 ml / min; serum phosphorus below 1.0 mg / dl (0.32 mmol / l).
* Patient with active viral infection (HBV, HCV and HIV), or uncontrolled acute infection.
* Patient with hypersensitivity to one of the active substances or to any of the excipients (non-medicinal ingredients).
* Patient with uncontrolled coagulation disorder, history of keloid scars
* Patient with an allergy to local anesthetics; any condition likely to interfere at the time of the pre-inclusion visit, with the evaluation of the main objective such as eczema, psychiatric disorders
* Patient with uncontrolled systemic parameters The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Percentage of patients no longer presenting S9.6:D5H6 RNA:DNA duplex | Day 0
  Biopsy screening for S9.6:D5H6 RNA:DNA duplex by immunofluorescence
Percentage of patients no longer presenting S9.6:D5H6 RNA:DNA duplex | Day 7
  Biopsy screening for S9.6:D5H6 RNA:DNA duplex by immunofluorescence

SECONDARY OUTCOMES:
Percentage change in endogenous reverse transcriptase | Day 0
  µUI/mL reverse transcriptase activity tested in serum assayed using CAVIDI HS Mg-RT kit
Percentage change in endogenous reverse transcriptase | Day 7
  µUI/mL reverse transcriptase activity tested in serum assayed using CAVIDI HS Mg-RT kit
Percentage change in Ki67 proliferation marker expression | Day 0
  Percentage of cells positive for Ki67 marker on cutaneous immunohistochemistry
Percentage change in Ki67 proliferation marker expression | Day 7
  Percentage of cells positive for Ki67 marker on cutaneous immunohistochemistry
Percentage change in CK10 differentiation marker expression | Day 0
  Percentage of cells positive for CK10 marker on cutaneous immunohistochemistry
Percentage change in CK10 differentiation marker expression | Day 7
  Percentage of cells positive for CK10 marker on cutaneous immunohistochemistry
Percentage change in filaggrin differentiation marker expression | Day 0
  Percentage of cells positive for filaggrin marker on cutaneous immunohistochemistry
Percentage change in filaggrin differentiation marker expression | Day 7
  Percentage of cells positive for filaggrin marker on cutaneous immunohistochemistry
Percentage change in CD4 inflammation marker expression | Day 0
  Percentage of cells positive for CD4 marker on cutaneous immunohistochemistry
Percentage change in CD4 inflammation marker expression | Day 7
  Percentage of cells positive for CD4 marker on cutaneous immunohistochemistry
Percentage change in CD8 inflammation marker expression | Day 0
  Percentage of cells positive for CD8 marker on cutaneous immunohistochemistry
Percentage change in CD8 inflammation marker expression | Day 7
  Percentage of cells positive for CD8 marker on cutaneous immunohistochemistry
Percentage change in CD11c inflammation marker expression | Day 0
  Percentage of cells positive for CD11c marker on cutaneous immunohistochemistry
Percentage change in CD11c inflammation marker expression | Day 7
  Percentage of cells positive for CD11c marker on cutaneous immunohistochemistry
Average percentage change of Psoriasis Area Severity Index | Day 7
  Scale of four variables of psoriasis severity (minimum score 0 maximum score 72)
Number of side effects | Day 7
  Anticipated side effects = diarrhea, vomiting, nausea, dizziness or headache, feeling weak or rash
Number of side effects | Day 14
  Anticipated side effects = diarrhea, vomiting, nausea, dizziness or headache, feeling weak or rash

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Stoebner, Principal Investigator — CHU Nimes
Locations (2):
- France (2):
  - CHU de Montpellier, Montpellier
  - CHU de Nimes, Nîmes